CLINICAL TRIAL: NCT03164720
Title: Serum/Urinary Monocyte Chemoattractant Protein-1 Level as a Marker for Lupus Nephritis
Brief Title: SSerum/Urinary Monocyte Chemoattractant Protein-1 Level as a Marker for Lupus Nephritis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rasha ahmed, assiut, Assiut University
Other Study IDs: assiut 8080
Record Dates: First submitted 2017-05-22; First posted 2017-05-24 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Systemic Lupus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Systemic lupus erythematosus (SLE) is a chronic inflammatory autoimmune disease affecting many organ systems. SLE includes a wide spectrum of severity, ranging from relatively mild manifestations (e.g. skin rash or non-erosive arthritis) to seriously disabling or even life threatening complications, such as lupus nephritis (LN) and neuropsychiatric disorders . LN is one of the most serious SLE complications since it is the major predictor of poor prognosis .

Lupus nephritis is a common major organ manifestation and main cause of morbidity and mortality of the disease . It is occurred in 30-50% of SLE patients at initial diagnosis and more prevalent in Asians and Blacks than other races . Approximately, 10-30% of LN patients will develop the end-stage renal disease (ESRD) within 15 years after diagnosis. The 5-year survival rate of a patient with severe LN is less than70-80%. Therefore, an involvement of renal disease activity is one of the most important prognostic factors for patients with SLE, and the diagnosis of SLE patients with LN has an important clinical implication in guiding the treatment of SLE in clinical settings.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a chronic inflammatory autoimmune disease affecting many organ systems. SLE includes a wide spectrum of severity, ranging from relatively mild manifestations (e.g. skin rash or non-erosive arthritis) to seriously disabling or even life threatening complications, such as lupus nephritis (LN) and neuropsychiatric disorders . LN is one of the most serious SLE complications since it is the major predictor of poor prognosis .

Lupus nephritis is a common major organ manifestation and main cause of morbidity and mortality of the disease. It is occurred in 30-50% of SLE patients at initial diagnosis and more prevalent in Asians and Blacks than other races . Approximately, 10-30% of LN patients will develop the end-stage renal disease (ESRD) within 15 years after diagnosis. The 5-year survival rate of a patient with severe LN is less than70-80% . Therefore, the diagnosis of SLE patients with LN has an important clinical implication in guiding the treatment of SLE in clinical settings.

Renal biopsies have remained the "gold standard" of assessing lupus nephritis (LN) patients not only at diagnosis but also to assess the efficacy of treatment. In contrast, current noninvasive laboratory markers for LN such as proteinuria, urine protein to creatinine ratio, creatinine clearance, antidsDNA, and complement levels are unsatisfactory because they lack sensitivity and specificity for differentiating renal activity and damage in LN.

The search for an accurate and reliable biomarker for lupus nephritis is particularly important since the only reliable method to evaluate it is by performing a kidney biopsy, that is an invasive procedure may not always be feasible. So significant effort has been put into identifying biomarkers that can anticipate impending lupus renal flare, forecast development of chronic kidney disease, or reflect kidney histology at time of flare .

Monocyte chemoattractant protein-1 (MCP1) is a chemokine that attracts monocytes/macrophages to sites of inflammation. MCP-1 is produced by mesangial, podocyte, and monocyte cells in response to various proinflammatory stimuli such as tumor necrosis factor alpha (TNF-

ELIGIBILITY:
Inclusion Criteria:

* revised American Collage of Rheumatology classification criteria for SLE

Exclusion Criteria:

* Patients with diabetes mellitus.
* patients with a diagnosis of overlap syndrome (coexistence of lupus with other connective tissue diseases such as rheumatoid arthritis or scleroderma)..
* Patients with urinary tract infection.
* Patients with end stage renal disease.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will include 60 patients with renal biopsy proven LN or without LN by laboratory investigation together with 20 healthy control age and sex matched with the patients.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Serum/Urinary monocyte chemoattractant protein-1 level as a marker for lupus nephritis | one year
  - Determine the levels of serum / urinary MCP-1 in patients with systemic lupus erythematosus

IPD SHARING:
Plan to Share IPD: Undecided
use Serum/Urinary monocyte chemoattractant protein-1 level as a marker for lupus nephritis